CLINICAL TRIAL: NCT05053035
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AL001 in C9orf72-Associated Amyotrophic Lateral Sclerosis
Brief Title: A Phase 2 Study to Evaluate AL001 in C9orf72-Associated ALS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor is considering a subsequent study in ALS, potentially with different inclusion/exclusion criteria.
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL001-ALS-201
Record Dates: First submitted 2021-09-01; First posted 2021-09-22 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AL001 (Experimental): AL001 every 4 weeks
  Interventions: Drug: AL001
- Placebo (Placebo Comparator): Placebo every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL001 — Administered via intravenous (IV) infusion
  Arms: AL001
Drug: Placebo — Administered via intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
A phase 2 double-blind, placebo-controlled study of AL001 in participants with C9orf72-associated ALS.

DETAILED DESCRIPTION:
This is a phase 2 double-blind, placebo-controlled trial to test the safety, tolerability, pharmacokinetics, and pharmacodynamics of AL001 in participants with C9orf72-associated Amyotrophic Lateral Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of C9orf72 mutation
* Diagnosis of ALS by revised El Escorial criteria
* Time since onset of muscle weakness due to ALS ≤36 months at the time of the Screening Visit
* Slow Vital Capacity (VC) ≥50% of predicted capacity at the time of the Screening Visit
* If taking riluzole, must be on a stable dose of riluzole for at least 30 days prior to the Screening Visit. Riluzole naive participants are allowed.
* If taking edaravone, must have completed at least one cycle of edaravone prior to the Screening Visit and plan to continue edaravone during the study. Edaravone naive participants are allowed.
* Females must not be pregnant, breastfeeding or planning to conceive within the study period. Males must agree to use acceptable contraception
* Capable of providing informed consent at the Screening visit and complying with study procedures throughout the study

Exclusion Criteria:

* Clinically significant, unstable, medical condition (other than ALS)
* Clinically significant heart disease, liver disease or kidney disease
* Cognitive impairment or dementia
* Current uncontrolled hypertension
* History of unresolved cancer
* Any experimental gene therapy
* Any experimental vaccine (any vaccine against COVID-19 either approved or administered under an Emergency Use Authorization is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Paganoni, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AL001 | Placebo
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL001 | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety and Tolerability of AL001 Measured by Number of Subjects With Adverse Events
Description: Count of participants with adverse events during the study treatment period
Time Frame: 24 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 2 | 2

2. Primary Outcome: Immunogenicity of AL001
Description: Count of participants positive for Anti-drug Antibodies (ADAs) to AL001 at week 24
Time Frame: Week 24
Population: Due to early termination of the study and insufficient sample size, no population-level analysis (within-group and between-group) was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

3. Primary Outcome: Pharmacokinetics (PK) of AL001 in Serum
Description: Concentration of AL001 in Serum at week 24
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 0
ng/mL | 705792.5 (87387.7916) |

4. Primary Outcome: Pharmacokinetics (PK) of AL001 in CSF
Description: Concentration of AL001 in Cerebrospinal fluid (CSF) at week 24
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 0
ng/mL | 547.5 (395.2727) |

5. Primary Outcome: Change From Baseline in Plasma Progranulin
Description: Evaluate the change from baseline to week 24 in plasma progranulin levels
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 2
ng/mL | 175 (2.8284) | -24.4 (9.3338)

6. Primary Outcome: Change From Baseline in CSF Progranulin
Description: Evaluate the change from baseline to week 24 in Cerebrospinal fluid (CSF) progranulin levels
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 2
ng/mL | 2.865 (1.0677) | -0.385 (0.3323)

7. Secondary Outcome: Change From Baseline in Plasma Neurofilament Light Chain
Description: Evaluate the change from baseline to week 24 in plasma neurofilament light chain levels
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 2
pg/mL | -0.35 (3.3234) | 1.9 (2.8284)

8. Secondary Outcome: Change From Baseline in CSF Neurofilament Light Chain
Description: Evaluate change from baseline to week 24 in Cerebrospinal fluid (CSF) neurofilament light chain levels
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AL001 | Placebo
Number analyzed (Participants) | 2 | 2
pg/mL | 995.5 (95.4594) | -1250.5 (825.1936)

ADVERSE EVENTS:
Time Frame: 32 Weeks
Arm/Group | AL001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL001 (N=3) | Placebo (N=2)
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Catheter site irritation (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Medical device site hemorrhage (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 1 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT05053035/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT05053035/SAP_001.pdf